CLINICAL TRIAL: NCT01207713
Title: Evaluation of the Functional and Cosmetic Outcome of Enucleation With Rectus End-to-end Suturing Surgical Technique in Coralline Hydroxyapatite Orbital Implants
Brief Title: A Modified Orbital Implantation Technique in Enucleation
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Jianan Wang, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: SAHZhejiangU
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Orbital Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — The investigators reviewed surgical records from July 2005 to March 2009, to identify patients who had received hydroxyapatite orbital implants after primary enucleation by a single surgeon
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the functional and cosmetic outcomes of enucleation with rectus end-to-end suturing surgical technique in hydroxyapatite orbital implants

DETAILED DESCRIPTION:
To assess the functional and cosmetic outcomes of enucleation with rectus end-to-end suturing surgical technique between 2005 and 2009. All the patients underwent primary enucleation and implantation of non-wrapped HA implants using a technique that involves drawing the ends of the rectus muscles anteriorly and suturing them into a cross-shape in front of the implant. Main outcome measures included occurrence of pain or discharge, soft tissue problems, implant motility, upper lid position, and patients' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

bilateral enucleation severely traumatized orbits, and little or no function of the extraocular muscles adjunctive radiotherapy and/or chemotherapy diabetes vessel inflammation follow-up of less than 6 months

Ages: 3 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who had received hydroxyapatite orbital implants after primary enucleation by a single surgeon from July 2005 to March 2009
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Ye, MD,Ph.D, Principal Investigator — second affiliated hospital,zhejiang university